CLINICAL TRIAL: NCT02506218
Title: Optimizing Meal and Snack Timing to Promote Health
Acronym: S43
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Professor Nutrition Science, Purdue University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1501015661
Record Dates: First submitted 2015-06-24; First posted 2015-07-23 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Dietary Modification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 10 + 20 g protein consumption (Experimental): 10 g breakfast followed by the consumption of a 20g whey protein shake
  Interventions: Dietary Supplement: 10 + 20 g protein consumption
- 30 g protein breakfast (Active Comparator)
  Interventions: Other: 30 g protein breakfast
- 10 g protein breakfast (Active Comparator)
  Interventions: Other: 10 g protein breakfast

INTERVENTIONS:
Dietary Supplement: 10 + 20 g protein consumption — whey isolate
  Arms: 10 + 20 g protein consumption
Other: 30 g protein breakfast — 30 g mixed meal breakfast
  Arms: 30 g protein breakfast
Other: 10 g protein breakfast — 10 g mixed meal breakfast
  Arms: 10 g protein breakfast

SUMMARY:
This study will be conducted using standardized techniques to collect blood samples via an acute, randomized, cross-over design. Subjects will be provided all of their meals the day prior to testing and participate in 3 testing days with a minimum of 1 week break between testing days and a maximum time commitment of 7 weeks. A trained phlebotomist will place a catheter and collect blood samples from an antecubital vein using sterile techniques.

ELIGIBILITY:
Inclusion Criteria:

25-39 years old

* BMI between 22-37 kg/m2
* Weight stable (± 4.5 kg) for the previous 3 months
* Not currently (or within the past 6 months) following a vigorous exercise regimen or weight loss program
* No acute illness
* Not smoking
* Not diabetic
* Not pregnant or planning pregnancy in the next 3 months
* Lactose tolerant
* Willing to limit purposeful activity for 48 hours prior to each testing day
* Willing to consume study foods and beverages.

Exclusion Criteria:

* <25 or >39 years old, BMI <22 or >37 kg/m2
* Currently (or within the past 6 months) following a vigorous exercise regimen greater than -3 - 45 minute exercise sessions per week
* Currently following a weight loss program where subject has lost greater than 4.5 kg
* Acute illness
* Smoking
* Diabetic
* Pregnant or planning pregnancy in the next 3 months
* Lactose intolerant
* Unwilling to consume study foods and beverages
* Peri and post-menopausal women.

Ages: 25 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Plasma amino acid concentration | 7 weeks
  Peak plasma concentration of amino acids

SECONDARY OUTCOMES:
Blood glucose concentration | 7 weeks
  Area under the curve of blood glucose

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States